CLINICAL TRIAL: NCT00145639
Title: Osteosarcoma 1999-A Study Of Intensive Chemotherapy Utilizing Ifosfamide, Carboplatin, and Doxorubicin for Adjuvant Chemotherapy for Treatment of Osteosarcoma
Brief Title: Osteosarcoma1999-A Study Of Intensive Chemotherapy for Osteosarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Immunex/Berlex (Industry); National Institutes of Health (NIH) (NIH)
Responsible Party: Fariba Navid, M.D., St.Jude Children's Research Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OS99
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2011-06

CONDITIONS: Osteosarcoma
Keywords: Osteosarcoma; Treatment, Carboplatin
MeSH Terms: conditions — Osteosarcoma | interventions — Ifosfamide; Carboplatin; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other)
  Interventions: Drug: Ifosfamide, Carboplatin, Doxorubicin; Procedure: Limb Sparing

INTERVENTIONS:
Drug: Ifosfamide, Carboplatin, Doxorubicin — See Detailed Description for treatment plan.
Procedure: Limb Sparing — See Detailed Description for treatment plan.

SUMMARY:
This trial (OS99) evaluates the use of ifosfamide, carboplatin, and doxorubicin in an up-front window before surgery for localized and resectable osteosarcoma. High-dose methotrexate, which may interfere with the dose-intensive delivery of other agents, is eliminated from the treatment of localized disease. The primary objective is to compare the response rate of pre-surgical chemotherapy comprised of ifosfamide, doxorubicin, and carboplatin to that obtained with ifosfamide and carboplatin in the St. Jude OS-91 trial for patients with non-metastatic resectable osteosarcoma. We hypothesize that the histologic response rate will be improved by the addition of one course of pre-operative chemotherapy on this trial compared to the previous OS-91 trial.

DETAILED DESCRIPTION:
This study has multiple research objectives:

* To compare the response rate of pre-surgical chemotherapy comprised of ifosfamide, doxorubicin, and carboplatin to that obtained with ifosfamide and carboplatin in the St. Jude OS-91 trial for patients with non-metastatic resectable osteosarcoma
* To continue the evaluation of dynamic contrast-enhanced magnetic resonance imaging (DEMRI) in predicting tumor response and accurately assessing the degree of response (continued from OS-91).
* To determine the feasibility of delivering outpatient-based chemotherapy for osteosarcoma using ifosfamide-doxorubicin-carboplatin.
* To determine whether resection of the primary site may be satisfactorily performed with a 3 cm margin of normal bone (rather than 5 cm).
* To study biologic and biochemical characteristics of the tumor cells that may be of prognostic significance
* To study the patients' and parents' perspectives of the patients' quality of life during and after treatment.

Description of Treatment Plan:

This study employs the following treatment strategy: neoadjuvant chemotherapy followed by definitive surgery for local control and adjuvant chemotherapy after tumor resection.

Pre-operative chemotherapy phase (weeks 0-12): Three courses of ifosfamide/carboplatin given every 3 weeks followed by one 3-week course of doxorubicin.Disease evaluation is performed after 3 courses and after 4 courses of chemotherapy.

Weeks 0, 3, and 6 - Ifosfamide-Carboplatin Ifosfamide: 2.65 gm/m2 IV daily over 15-30 minutes x 3 (Days 1, 2, 3) with MESNA. Carboplatin: dose based on GFR and targeted to an AUC of 8 mg/mL/min, given IV over 1 hour (Day 1 only)

Week 9- Evaluation, followed by Doxorubicin Doxorubicin: 25 mg/m2 IV over 1 hour, daily x 3

Week 12 Evaluation followed by definitive Surgery Local control by amputation or limb-salvage procedure

Post-operative chemotherapy (Weeks 14-35) Ifosfamide, carboplatin, and doxorubicin in two-agent pairs for approximately 35 weeks.

Week 14 - Ifosfamide-Doxorubicin Ifosfamide: 2.65 gm/m2 IV daily over 15-30 minutes x 3 (Days 1, 2, 3) with MESNA, Doxorubicin: 25 mg/m2 IV over 1 hour, daily x 2 (Days 1 and 2)

Week 17 - Ifosfamide-Carboplatin Ifosfamide: 2.65 gm/m2 IV daily over 15-30 minutes x 3 (Days 1, 2, 3) with MESNA, Carboplatin: targeted to an AUC of 8 mg/mL/min given IV over 1 hour (Day 1 only)

Week 20 - Carboplatin-Doxorubicin Carboplatin: targeted to an AUC of 8 mg/mL/min given IV over 1 hour (Day 1 only), Doxorubicin: 25 mg/m2 IV over 1 hour, daily x 2 (Days 1 and 2)

Week 23 - Evaluation, followed by Ifosfamide:

Doxorubicin. Ifosfamide: 2.65 gm/m2 IV daily over 15-30 minutes x 3 (Days 1, 2, 3) with MESNA, Doxorubicin: 25 mg/m2 IV over 1 hour, daily x 2 (Days 1 and 2)

Week 26 - Ifosfamide-Carboplatin Ifosfamide: 2.65 gm/m2 IV daily over 15-30 minutes x 3 (Days 1, 2, 3) with MESNA, Carboplatin: targeted to an AUC of 8 mg/mL/min given IV over 1 hour (Day 1 only)

Week 29 - Carboplatin-Doxorubicin Carboplatin: targeted to an AUC of 8 mg/mL/min given IV over 1 hour (Day 1 only), Doxorubicin: 25 mg/m2 IV over 1 hour, daily x 2 (Days 1 and 2)

Week 32 - Evaluation, followed by Ifosfamide-Doxorubicin. Ifosfamide: 2.65 gm/m2 IV daily over 15-30 minutes x 3 (Days 1, 2, 3) with MESNA, Doxorubicin: 25 mg/m2 IV over 1 hour, daily x 2 (Days 1 and 2)

Week 35 - Carboplatin-Doxorubicin Carboplatin: targeted to an AUC of 8 mg/mL/min given IV over 1 hour (Day 1 only), Doxorubicin: 25 mg/m2 IV over 1 hour, daily x 2 (Days 1 and 2)

ELIGIBILITY:
Inclusion Criteria:

* All subjects with histologically proven high-grade osteosarcoma,chondrosarcoma, MFH, fibrosarcoma or chondrosarcoma of bone, whose tumors are potentially resectable (either by limb sparing, en bloc resection, or amputation) and have no evidence of metastasis.
* Adequate liver, renal and cardiac function.
* Age: Younger than 25 years old

Exclusion Criteria:

* Prior chemotherapy

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 1999-05; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Histologic response rate | After all patients have undergone definitive surgery and become evaluable for histologic response evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Fariba Navid, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (4):
- United States (3):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Washington University Medical Center, St Louis, Missouri
  - St.Jude Children's Research Hospital, Memphis, Tennessee
- Hospital Luis Calvo Mackenna, Santiago, Chile

REFERENCES:
- [Background] Crews KR, Stewart CF, Liu T, Rodriguez-Galindo C, Santana VM, Daw NC. Effect of fractionated ifosfamide on the pharmacokinetics of irinotecan in pediatric patients with osteosarcoma. J Pediatr Hematol Oncol. 2004 Nov;26(11):764-7. doi: 10.1097/00043426-200411000-00016. PMID 15543015
- [Background] Sanders RP, Drissi R, Billups CA, Daw NC, Valentine MB, Dome JS. Telomerase expression predicts unfavorable outcome in osteosarcoma. J Clin Oncol. 2004 Sep 15;22(18):3790-7. doi: 10.1200/JCO.2004.03.043. PMID 15365076
- [Background] McCarville MB, Barton EH, Cameron JR, Xiong X, Daw NC, Kaste SC, Wu S, Glass JO, Reddick WE. The cause and clinical significance of central tumor photopenia on thallium scintigraphy of pediatric osteosarcoma of the extremity. AJR Am J Roentgenol. 2007 Feb;188(2):572-8. doi: 10.2214/AJR.06.0292. PMID 17242270
- [Background] Freeman SS, Allen SW, Ganti R, Wu J, Ma J, Su X, Neale G, Dalton J, Billups C, Dome JS, Daw NC, Khoury JD. Osteosarcoma tumors commonly express EGFR and harbor frequent gains at the EGFR locus and losses at the PTEN Locus. Clin Cancer Res (Submitted).
- [Background] Rivera GK, Quintana J, Villarroel M, Santana VM, Rodriguez-Galindo C, Neel MD, Velez G, Ribeiro RC, Daw NC. Transfer of complex frontline anticancer therapy to a developing country: the St. Jude osteosarcoma experience in Chile. Pediatr Blood Cancer. 2008 Jun;50(6):1143-6. doi: 10.1002/pbc.21444. PMID 18085687
- [Background] McCarville MB, Romano E, Daw N, Xiong X, Reddick W, Kaste S. Etiology of the 201Thallium
- [Background] McCarville MB, Reddick WE, Xiong X, Kaste SC, Daw NC. Clinical significance of the 201Thallium donut-sign in primary extremity osteosarcoma. Presented at the 2006 Society of Pediatric Radiology and European Society of Paediatric Radiology's Fifth Conjoint Meeting, Montreal, Quebec, Canada, May 18-20, 2006.
- [Background] Kaste SC, Waszilycsak G, McCarville MB, Daw NC. Excess cancer mortality in pediatric thallium imaging. Presented at the 2006 Society of Pediatric Radiology and European Society of Paediatric Radiology's Fifth Conjoint Meeting, Montreal, Quebec, Canada, May 18-20, 2006.
- [Background] Freeman SS, Allen SW, Ganti R, Wu J, Ma J, Su X, Neale GA, Dalton JD, Billups CA, Dome JS, Daw NC, Khoury JD. EGFR expression and copy number gain are common in osteosarcoma. Presented at the US and Canadian Academy of Pathology Annual Meeting, San Diego, California, March 24-30, 2007.
- [Background] Reddick WE, Hoffer FA, Billups CA, Jenkins JJ, Wu J, Daw NC. Response assessment using dynamic MR imaging in non-metastatic osteosarcoma. To be presented at the ASCO Annual Meeting, Chicago, Illinois, June 2007.
- [Background] Rivera GK, Quintana J, Villarroel M, Rodríguez C, Santana VM, Ribeiro RC, Daw NC. Conduct of an international collaborative osteosarcoma trial at centers in a developed and developing country. To be presented at the ASCO Annual Meeting, Chicago, Illinois, June 2007.
- See also: St. Jude Children's Research Hospital — http://www.stjude.org